CLINICAL TRIAL: NCT03702959
Title: Antenatal Betamethasone and the Risk of Neonatal Hypoglycemia: It's All About Timing
Brief Title: Antenatal Betamethasone and the Risk of Neonatal Hypoglycemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Yaniv Zipori MD, Principal Investigator, Rambam Health Care Campus
Other Study IDs: 0205 - 18 - RMB
Record Dates: First submitted 2018-10-08; First posted 2018-10-11 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Hypoglycemia
MeSH Terms: conditions — Hypoglycemia | interventions — Betamethasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Betamethasone group 1: Betamethasone Group 1 (5am-11am)
  Interventions: Drug: Betamethasone
- Betamethasone Group 2: Betamethasone Group 2 (11am-5pm)
  Interventions: Drug: Betamethasone
- Betamethasone Group 3: Betamethasone Group 3 (5pm-11pm)
  Interventions: Drug: Betamethasone
- Betamethasone Group 4: Betamethasone Group 4 (11pm-5am).
  Interventions: Drug: Betamethasone

INTERVENTIONS:
Drug: Betamethasone — Corticosteroids

SUMMARY:
A single "supraphysiological" course of exogenous corticosteroids is recommended between 24-34 weeks' gestation to minimize the adverse sequelae associated with prematurity. The 24-hour profile of endogenous corticosteroids normally follows a diurnal rhythm with the highest serum level occurs between 5am-11am and nadir over 12 hours.

DETAILED DESCRIPTION:
A retrospective study from January 2010 to December 2017. Eligible for analysis are: singleton pregnancies between 24 - 34 weeks' gestation who were given a single course of intramuscular betamethasone. Single course comprised of two separate doses of 12 mg given 24 hours apart. Each woman was allocated into one of the four pre-defined groups based on the time the intramuscular betamethasone was administered; Group 1 (5am-11am), group 2 (11am-5pm), group 3 (5pm-11pm) and group 4 (11pm-5am). The investigators hypothesized that exogenous corticosteroids given during the nadir state of endogenous corticosteroids activity could alter maternal and fetal glucose homeostasis.

ELIGIBILITY:
Inclusion Criteria:

• women between 24 - 34 weeks' gestation who were admitted and given a single course of intramuscular betamethasone for threatened preterm labor in our institution

Exclusion Criteria:

* higher order multiple pregnancies
* women who were given more than one course of betamethasone during the course of the current pregnancy
* known major congenital anomalies.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women and their newborns
Study Population: This is a retrospective study at Rambam Health Care Campus.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of neonatal hypoglycemia | 7 years
  Incidence of neonatal hypoglycemia, glucose ˂ 40 mg/dL at any time

CONTACTS AND LOCATIONS:
Overall Officials: Yaniv Zipori, M.D, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided
The study is expected to be published after completion